CLINICAL TRIAL: NCT07287618
Title: Clinical Evaluation of Potassium and Ionized Calcium Tests Using the i-STAT CG8+ Cartridge With the i-STAT 1 Analyzer for Capillary Specimens
Brief Title: Evaluation of Potassium (K) and Ionized Calcium (iCa) Tests Using Capillary Specimens
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Point of Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CS-2025-0001
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hematologic Tests
Keywords: Potassium (K) ionized calcium (iCa)
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Method Comparison Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Method comparison for K and iCa tests using capillary whole blood specimens. (Other): Performance comparison: Using results from capillary whole blood specimens collected from fingerstick(s) from each subject enrolled in the study, the performance between i-STAT potassium (K) and ionized calcium (iCa) tests using i-STAT CG8+ cartridge on i-STAT 1 analyzer and a comparator blood analysis system will be compared.
  Interventions: Diagnostic Test: Blood draw

INTERVENTIONS:
Diagnostic Test: Blood draw — Capillary whole blood specimens collected from fingerstick(s) from each enrolled subject using blood collection capillary tubes.

SUMMARY:
The objective of this study is to compare the performance of blood tests using the i-STAT 1 System against a comparator blood analysis system.

DETAILED DESCRIPTION:
To compare the performance of the i-STAT potassium (K) and ionized calcium (iCa) tests using the i-STAT CG8+ cartridge on the i-STAT 1 analyzer to the performance of K and iCa tests on a comparator blood analysis system using results from two separate capillary specimens from each subject enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated consent form (waiver/alteration of consent, waiver of documentation of consent may be acceptable, per IRB)
2. ≥ 18 years of age

Exclusion Criteria:

1. Previous enrollment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 425 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Method Comparison for potassium (K) and ionized calcium (iCa) blood tests. | Thirty (30) minutes from subject enrollment to the end of the blood draw and testing.
  Specimen testing of K and iCa in mmol/L will be performed using the i-STAT CG8+ cartridge on the i-STAT analyzer and a comparator blood analysis system with prospectively collected capillary specimens.
  Subjects with one valid capillary result on the i-STAT CG8+ cartridge and one valid result on the comparator blood analysis system will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Manish Gupta, MS, MBA, Study Director — Abbott Point of Care
Locations (3):
- United States (3):
  - University of New Mexico, Albuquerque, New Mexico
  - Penn State Health Milton S. Hershey Medical Center (Hershey), Hershey, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No